CLINICAL TRIAL: NCT03059485
Title: A Randomized Phase II Clinical Trial of Dendritic Cell/AML Fusion Cell Vaccine Versus Observation in Patients Who Achieve a Chemotherapy-induced Remission
Brief Title: DC/AML Fusion Cell Vaccine vs Observation in Patients Who Achieve a Chemotherapy-induced Remission
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Celgene (Industry); Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Jacalyn Rosenblatt, Jacalyn Rosenblatt, MD, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-593
Record Dates: First submitted 2017-02-15; First posted 2017-02-23 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Acute Myelogenous Leukemia
Keywords: Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia | interventions — Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DC/AML Vaccine (Experimental): - Patients will be vaccinated with DC/AML Fusion Vaccine
  Interventions: Biological: DC/AML Fusion Vaccine; Other: Observation
- Observation (Experimental): - Patients will be monitored with routine labs and bone marrow biopsies
  Interventions: Other: Observation

INTERVENTIONS:
Biological: DC/AML Fusion Vaccine — The Dendritic Cell Fusion Vaccine is an investigational agent that tries to help the immune system to recognize and fight against cancer cells
  Arms: DC/AML Vaccine
Other: Observation — Traditional care provided by the hospital.

SUMMARY:
This research study is studying a cancer vaccine called Dendritic Cell/AML Fusion vaccine (DC/AML vaccine) as a possible treatment for Acute Myelogenous Leukemia (AML).

The interventions involved in this study are:

-Dendritic Cell/AML Fusion vaccine (DC/AML vaccine)

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational intervention to learn whether the intervention works in treating a specific disease. "Investigational" means that the intervention is being studied.

The FDA (the U.S. Food and Drug Administration) has not approved the DC/AML vaccine as a treatment for any disease.

The FDA (the U.S. Food and Drug Administration) has not approved durvalumab as a treatment for AML.

In this research study, the investigators are determining if the DC/AML vaccine can be used safely in subjects with acute leukemia after finishing chemotherapy, and whether the DC/AML vaccine is capable of producing immune responses against leukemia alone. Cancer cells are foreign to the body and have unique markers that distinguish them from normal cells. These markers can potentially serve as targets for the immune system. An immune response is any reaction by the immune system; a complex system that is responsible for distinguishing us from everything foreign to us, and for protecting us against infections and foreign substances.

The Dendritic Cell Fusion Vaccine is an investigational agent that tries to help the immune system to recognize and fight against cancer cells. Unlike a standard vaccine that is used to prevent infections, cancer vaccines are being studied to see if they can fight cancers that are already in the body. Laboratory studies have shown that when dendritic cells and tumor cells are brought together, the dendritic cells can stimulate immune responses against the tumor and, in some cases, cause the tumor to shrink.

ELIGIBILITY:
Step 1: Eligibility Criteria for Tumor Collection

Inclusion Criteria

* Patients must have AML at initial diagnosis or at first relapse
* Patients must be ≥ 55 years old
* ECOG performance status ≤2 (Appendix A)
* Patients must have normal organ and marrow function as defined below:

total bilirubin ≤ 2.0 mg/dL AST(SGOT)/ALT(SGPT) ≤3 × institutional upper limit of normal creatinine ≤ 2.0 mg/dl

* The effects of DC/AML fusion cells on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria

-Active or prior documented autoimmune or inflammatory disorders including but not limited to the following:

--GI Disorders: (including inflammatory bowel disease [eg, ulcerative colitis, Crohn's disease], diverticulitis (with the exception of a prior episode that has resolved), celiac disease, or other serious gastrointestinal chronic conditions associated with diarrhea.

* Systemic lupus erythematosus
* Wegener's syndrome [granulomatosis with polyangiitis]
* Myasthenia gravis
* Graves' disease
* Rheumatoid arthritis
* Hypophysitis
* Uveitis

The following are exceptions to this criterion: subjects with vitiligo or alopecia; subjects with hypothyroidism (eg, following Hashimoto syndrome) stable on hormone replacement; or subjects with psoriasis not requiring systemic treatment..

* Because of compromised cellular immunity, patients who have a Known human immunodeficiency virus (HIV), hepatitis C virus (HCV) or evidence of active hepatitis B virus (HBV).
* Patients must not have significant cardiac disease characterized by symptomatic congestive heart failure, unstable angina pectoris, clinically significant cardiac arrhythmia
* Patients must not be pregnant. All premenopausal patients will undergo pregnancy testing. Men will agree to not father a child while on protocol treatment. Men and women will practice effective birth control while receiving protocol treatment.
* Individuals with a history of a different malignancy are ineligible except for the following circumstances. Individuals with a history of other malignancies are eligible if they have been disease-free for at least 5 years and are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancers are eligible if diagnosed and treated within the past 5 years: non-invasive cancer (such as, any in situ cancers) and basal cell or squamous cell carcinoma of the skin.
* Prior allogeneic transplant

Step 2: Eligibility Criteria Prior to Randomization

Inclusion Criteria

* Patients must have obtained a complete remission with chemotherapy defined by the absence of circulating blasts, and less than 5% blasts on bone marrow examination following hematopoietic recovery
* Patient required no more than 2 cycles of chemotherapy or 4 cycles of a hypomethylating agent (alone or in conjunction with venetoclax) to achieve remission.
* Resolution of all chemotherapy related grade III-IV toxicity as per CTC criteria 4.0
* Laboratories:

Absolute Neutrophil Count >1,000/uL Platelets > 50,000/uL Bilirubin < 2.0 mg/dL Creatinine <2.0 mg/dL AST/ALT < 3.0 x ULN

- For patients with evidence of minimal residual disease prior to vaccination, assessment of minimal residual disease status by cytogenetics or FISH will be followed post vaccination.

Exclusion Criteria

* Patients must not have serious intercurrent illness such as infection requiring IV antibiotics, or significant cardiac disease characterized by significant arrhythmia, ischemic coronary disease or congestive heart failure
* Patients who, with their treating physician, choose to proceed with an allogeneic transplant at the time of remission will not be eligible for randomization
* Active or prior documented autoimmune or inflammatory disorders including but not limited to the following:

  * GI Disorders: (including inflammatory bowel disease [eg, ulcerative colitis, Crohn's disease], diverticulitis (with the exception of a prior episode that has resolved), celiac disease, or other serious gastrointestinal chronic conditions associated with diarrhea.

    * Systemic lupus erythematosus
    * Wegener's syndrome [granulomatosis with polyangiitis]
    * Myasthenia gravis
    * Graves' disease
    * Rheumatoid arthritis
    * Hypophysitis
    * Uveitis

The following are exceptions to this criterion: subjects with vitiligo or alopecia; subjects with hypothyroidism (eg, following Hashimoto syndrome) stable on hormone replacement; or subjects with psoriasis not requiring systemic treatment.

* Current or prior use of immunosuppressive medication within 14 days prior to first dose of vaccine. The following are exceptions to this criterion: intranasal, inhaled, topical or local steroid injections (eg. intra-articular injection); steroids as premedication for hypersensitivity reactions; systemic corticosteroid at physiologic doses not to exceed 10mg/day of prednisone or equivalent
* Known human immunodeficiency virus (HIV), hepatitis C virus (HCV) or evidence of active hepatitis B virus (HBV).
* History of hypersensitivity to durvalumab or any excipient
* Receipt of live attenuated vaccination within 30 days prior the first vaccine
* Female subjects who are pregnant, breast-feeding or female patients of reproductive potential who are not employing an effective method of birth control from starting vaccine, including dosing interruptions through 90 days after receipt of the last vaccine. Refrain from egg cell donation during vaccination and for at least 90 days after the last vaccine.
* Male subjects who are not employing an effective method of birth control from starting vaccine, including dosing interruptions through 90 days after receipt of the last vaccine. Refrain from sperm donation during vaccination and for at least 90 days after the last vaccine.

Step 3: Eligibility Criteria Prior to Treatment or Observation

* Resolution of all chemotherapy related grade III-IV toxicity as per CTC criteria 4.0
* Laboratories:

WBC > 2.0 X 103/uL Platelets > 50,000/uL Bilirubin < 2.0 mg/dL Creatinine <2.0 mg/dL AST/ALT < 3.0 x ULN

- At least 2 doses of fusion vaccine were produced (Arm A only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2026-09-04 (Estimated); Study Completion 2026-12-04 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 2 years

SECONDARY OUTCOMES:
Overall Survival | 2 years
Assessing Toxicity using CTCAE version 4.03 | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jacalyn Rosenblatt, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (4):
- United States (4):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No